CLINICAL TRIAL: NCT00505479
Title: Iodine Status in Pregnant Women and Their Newborns: is Congenital Hypothyroidism Related to Iodine Deficiency in Pregnancy?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Other Study IDs: G20020584
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Congenital Hypothyroidism; Pregnancy; Iodine Deficiency
Keywords: Congenital Hypothyroidism; pregnancy; iodine; deficiency
MeSH Terms: conditions — Congenital Hypothyroidism

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Iodine is an essential component of thyroid hormone, which is necessary for many metabolic processes as well as the maturation of the CNS. Deficiencies of iodine have deleterious effects on both pregnant women and infants. The iodine status of the population after implementation of the universal salt iodization program in Zhejiang province has not been known. This study was to determine whether pregnant women show evidence of iodine deficiency, and to examine the correlation between maternal urine iodine concentration and newborn thyroid function.

DETAILED DESCRIPTION:
Iodine is an essential component of thyroid hormone, which is necessary for many metabolic processes as well as the maturation of the CNS. Deficiencies of iodine have deleterious effects on both pregnant women and infants. The iodine status of the population after implementation of the universal salt iodization program in Zhejiang province has not been known. This study was to determine whether pregnant women show evidence of iodine deficiency, and to examine the correlation between maternal urine iodine concentration and newborn thyroid function.

Healthy women at 12 weeks' gestation and over from four different areas in Zhejiang province were enrolled to participate this program from May 2007 to May 2010. Women consented to provide urine samples and salt samples during pregnancy (12, 16, 24 weeks' gestation and before delivery), and give permission to access their newborn's TSH value. Urinary iodine concentration (UIC) was determined by ammonium persulfate digestion microplate method, and TSH was determined by a time resolved fluoro-immunoassay (TRFIA). The diagnostic standard for congenital hypothyroidism was: TSH ≥ 20 mU/L and declined FT4 levels. Compare the correlation to effects with different level of iodine content in salt, maternal UIC and neonatal TSH. Investigate the optimal level of iodine content in salt in different areas in ZheJiang province.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in Zhejiang province (and their newborns)

Exclusion Criteria:

* Endocrine disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-05; Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: zhengyan Zhao, M.D., Study Director — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China